CLINICAL TRIAL: NCT00987922
Title: Mild Hypothermia in Acute Ischemic Stroke After Thrombolytic Therapy: a Prospective,Open,Randomized,Single-center,Safety and Feasibility Study
Brief Title: Mild Hypothermia in Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Katja Piironen, MD, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FI-HUCH-220424
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Brain Ischemia
Keywords: Stroke; Acute; Infarction; Ischemic; Thrombolysis; Mild; Hypothermia
MeSH Terms: conditions — Brain Ischemia; Stroke; Infarction; Ischemia; Lymphoma, Follicular; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypothermia (Experimental)
  Interventions: Device: Hypothermia
- Control (No Intervention)

INTERVENTIONS:
Device: Hypothermia — Hypothermia to core temperature of 35C for 12 hours, rewarming rate 0.2C until the patient reaches 36.8C
  Arms: Hypothermia

SUMMARY:
Hypothesis: Mild hypothermia using non-invasive temperature management system in a stroke unit is safe and feasible in spontaneously breathing, alteplase-thrombolyzed patients with acute ischemic stroke.

DETAILED DESCRIPTION:
Fever is associated with higher stroke mortality and poor outcome, but it is yet unknown whether this association is causative or epiphenomenal.

In temporary brain ischemia rodent models hypothermia results in a significant increase in the number of surviving neurons and smaller infarction size as measured with histological examination after death.

Therapeutic effect has been shown in clinical trials in comatose cardiac arrest patients and newborn infants with perinatal hypoxic-ischemic brain injury.

Design: A prospective, open, randomized single-center study.

Study population: 36 patients, 18-85 years of age presenting with symptoms of acute ischemic hemispheric stroke with persisting significant neurological deficit (NIHSS 7-20 or NIHSS 2 for dysphasia or NIHSS 3 for paralysis of upper or lower limb) at 2 hours after thrombolysis.

Method: Patients are randomized to hypothermia- or control-group via randomization envelopes. Patients assigned to receive hypothermia are cooled to a core temperature of 35°C for 12 hours by means of a non-invasive temperature management system and cold i.v. fluids. Induction of hypothermia is initiated within 6 hours of symptom onset. After 12 hours of successful cooling the target temperature is gradually raised to achieve slow re-warming of 0.2°C/h until the core temperature reaches 36.8°C.

Patients are breathing spontaneously and shivering is controlled with following medication; dexmedetomidine 0.2-0.7 µg/kg/h (i.v.), buspirone 5-20 mg x 3 (nasogastric tube), and meperidine 25mg (i.v.) when needed.

Core temperature, blood pressure (BP), oxygen saturation, ECG and EEG are measured continuously and registered hourly. Blood tests will be taken before, during and after hypothermia. Brain CT will be controlled when normothermia is reached, no later than 30 hours from symptom onset. Brain MRI will be performed 3-7 days from symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic hemispheric stroke treated with Actilyse(tPA)-thrombolysis according to Meilahti protocol
* NIHSS 7-20 (after thrombolysis) or a significant paresis of arm or leg (NIHSS 3, no movement against gravity) or a significant dysphasia (NIHSS 2-3) despite of the total NIHSS score
* Symptom onset within 6 hour

Exclusion Criteria:

* Platelet count < 75,000/mm3
* Known coagulopathy (INR spontaneously >1.5)
* Hemodynamical unstability
* Recent history of angina pectoris or acute myocardial infarction
* Sepsis within 72 hours
* Pregnancy
* Pre-existing neurological disability with modified Rankin Scale Score>2
* Known allergy or intolerance to buspirone, dexmedetomidine, meperidine
* Intracranial hemorrhage in brain CT scan
* Intracranial mass lesion (i.e., abscess, tumor, or infection)
* Participation in an other therapy trial within last 3 months
* Hypothermia- treatment cannot be initiated within 6 hours of symptom onset
* Protocol violation in thrombolytic therapy
* Any condition where researchers assume that the patient is not suitable (must be reasoned)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The proportion of patients maintaining temperature below 36.0°C 80% of the 12-hour hypothermia period. | 12 hours

SECONDARY OUTCOMES:
The incidence of intracerebral hemorrhage, infections, hemodynamically significant cardiac arrhythmias, severe disturbance of electrolytes and fluid balance, thrombocytopenia, and serious adverse events | 14 days
All-cause mortality during acute phase (7 days), 1 month, and 3 month follow-up; and readmission to hospital for any reason within 3-months. | 3 months
The proportion of modified Rankin Scale-responders (mRS 0-2), Barthel Index, NIHSS, Glasgow Outcome Scale | 3 months
Neuropsychological tests | 3 months
Size of infarction in MRI, and grading of the possible hemorrhagic transformation according to SITS scale (MRI includes scout images, DWI, T1, T2, FLAIR, T2*, and MR angiography) | 3-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Markku Kaste, MD, PhD, Principal Investigator — Helsinki University Central Hospital

REFERENCES:
- [Derived] Piironen K, Tiainen M, Mustanoja S, Kaukonen KM, Meretoja A, Tatlisumak T, Kaste M. Mild hypothermia after intravenous thrombolysis in patients with acute stroke: a randomized controlled trial. Stroke. 2014 Feb;45(2):486-91. doi: 10.1161/STROKEAHA.113.003180. Epub 2014 Jan 16. PMID 24436240